CLINICAL TRIAL: NCT03756610
Title: Transcranial Alternating Current Stimulation (tACS) for Cognitive Impairments in Patients With Schizophrenia: a Randomized Controlled Trial
Brief Title: Transcranial Alternating Current Stimulation (tACS) for Cognitive Impairments in Patients With Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-24
Record Dates: First submitted 2018-10-27; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-10

CONDITIONS: Schizophrenia
Keywords: tACS; schizophrenia; cognition; fMRI
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active tACS & active boosting group (Active Comparator): The active tACS & active boosting group will be stimulated with 10 sessions of active alternating current stimulation (tACS) and 5 booster sessions of active tACS.
  Interventions: Device: Active tACS; Device: Active boosting
- Active tACS & sham boosting group (Other): The active tACS & sham boosting group will be stimulated with 10 sessions of active alternating current stimulation (tACS) and 5 booster sessions of sham tACS.
  Interventions: Device: Active tACS; Device: Sham boosting
- Sham tACS & sham boosting group (Sham Comparator): The sham tACS & sham boosting group will be stimulated with 10 sessions of sham alternating current stimulation (tACS) and 5 booster sessions of sham tACS.
  Interventions: Device: Sham tACS; Device: Sham boosting

INTERVENTIONS:
Device: Active tACS — Placement of stimuli electrodes will be: a) active electrode over the left DLPFC (F3), and b) reference electrode over the right parietal region (P2). The exact location of electrodes will be determined by the 10/20 EEG method with EEG cap. Subjects will have tACS sessions on consecutive days (weekends and holidays excluded). Each subject will have 10 active tACS sessions.The active tACS group will be stimulated with a 2 mA current for 20 minutes.
  Arms: Active tACS & active boosting group; Active tACS & sham boosting group
Device: Sham tACS — Placement of stimuli electrodes will be: a) active electrode over the left DLPFC (F3), and b) reference electrode over the right parietal region (P2). The exact location of electrodes will be determined by the 10/20 EEG method with EEG cap. Subjects will have tACS sessions on consecutive days (weekends and holidays excluded). Each subject will have 10 sham tACS sessions.The sham tACS group will have stimulation lasting only 40 seconds though the electrodes will remain in place for 20 min.
  Arms: Sham tACS & sham boosting group
Device: Active boosting — Placement of stimuli electrodes will be: a) active electrode over the left DLPFC (F3), and b) reference electrode over the right parietal region (P2). The exact location of electrodes will be determined by the 10/20 EEG method with EEG cap. Subjects will have tACS sessions on consecutive days (weekends and holidays excluded).One month later after initial treatment, each subject will have 5 booster sessions of active tACS.The active boosting group will be stimulated with a 2 mA current for 20 minutes.
  Arms: Active tACS & active boosting group
Device: Sham boosting — Placement of stimuli electrodes will be: a) active electrode over the left DLPFC (F3), and b) reference electrode over the right parietal region (P2). The exact location of electrodes will be determined by the 10/20 EEG method with EEG cap. Subjects will have tACS sessions on consecutive days (weekends and holidays excluded).One month later after initial treatment, each subject will have 5 booster sessions of sham tACS.The sham boosting group will have stimulation lasting only 40 seconds though the electrodes will remain in place for 20 min.
  Arms: Active tACS & sham boosting group; Sham tACS & sham boosting group

SUMMARY:
This trial attempts to investigate whether 10 sessions of tACS improves cognitive function, especially which domains of cognitive function are most improved and to investigate whether 10 sessions of tACS affecting brain activation during a working memory task and changes patterns of brain connectivity networks.Subjects will be divided into 2 groups 2:1, active and sham tACS. 50 subjects will be in the active group, and 25 subjects in the sham group (specific numbers to be decided on later).

DETAILED DESCRIPTION:
Schizophrenia patients (SZ) show profound and persistent cognitive deficits in attention, executive processing, and verbal and visuospatial memory, which persist even after psychotic symptoms are ameliorated. Cognitive deficits may be more important in preventing functional, occupational, and social recovery in SZ than other symptom domains and are not effectively treated by current pharmacological approaches. Alternating current stimulation (tACS) is less expensive than other modalities (e.g. repetitive transcranial magnetic stimulation; rTMS), easily available, and has a good safety profile in healthy controls (HC) and SZ. The ability to entrain γ oscillations with 40Hz tACS, might compensate more specifically for this deficit in γ oscillations in schizophrenia, and, may therefore, produce more robust behavioral improvements in working memory and other aspects of cognition.However, no studies have looked at the effects of multiple daily tACS stimulation at a 40HZ γ frequency on cognitive function and symptoms in schizophrenia. This provides a rationale for the current study, which proposes to investigate the effects of 10 sessions of 40HZ tACS on cognitive functions, symptoms in schizophrenia.

Active vs. sham treatment will be randomly assigned in a 2:1 fashion (A:S) in groups using computer generated lists. Subjects and tDCS testers or evaluators will be blind to treatment. Subjects will be evaluated with cognitive, symptom and functional measures at baseline, within 1 day ( or 2 days fro some measures) after 10 sessions, 2 weeks after 10 sessions, 1 month after 10 sessions, and 2 months after 10 sessions.After the 1 month evaluation, subjects in the initial active tACS group will be randomly assigned to receive either 5 booster sessions of either active or sham tACS ( 25 subjects each), following parameters used in the initial treatment. Subjects in the initial Sham group will receive 5 booster session Sham tACS. Participants will be scanned once prior to tACS sessions, and within 3 days after the 10th tACS session, using our Siemens 3T Tim Verio MRI scanner with a standard 32-channel phased-array head coil.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have cognitive deficits as indicated by a score of < 85 on RBANS, and meet criteria for DSM-5 diagnosis of chronic SZ, schizoaffective disorder (SA), or schizophreniform disorder (SZF), and who are stably treated with antipsychotic medications and are not in acute exacerbation of illness symptoms.

Exclusion Criteria:

* Patients with risk factors for an MRI scan, seizure disorder, and for women of childbearing age who are pregnant or regularly engaging in sexual activity and not regularly using an acceptable birth control method (systemic or double-barrier).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
changes in The MATRICS Consensus Cognitive Battery (MCCB) | Change from Baseline MCCB at 2 weeks.
changes in Neuroimage changes in Magnetic Resonance Imaging (MRI) | Change from Baseline at 2 weeks.
  Including T1, resting state functional MRI, task based functional MRI and Diffusion Tensor Imaging(DTI)
changes in Gamma oscillation intensity ( 40-80 Hz) over the left and right frontal lobe | Change from Baseline at 2 weeks.
  measured by electroencephalogram (EEG)

SECONDARY OUTCOMES:
N-back task | At baseline,1-week, 2-week, 4-week, and 8-week follow-up.
  to test working memory
The Paced Auditory Serial Addition Task (PASAT) | At baseline,2-week, 4-week, and 8-week follow-up.
  to test Verbal Working memory
The Positive and Negative Syndrome Scale (PANSS) | At baseline,2-week, 4-week, and 8-week follow-up.
  PANSS was assessed using 30 basic items to form three subscales: positive, negative, and general psychopathological scales.The value of each item is ranging from 1 to 7, higher values represent more serious symptoms of schizophrenia.
The USCD Performance- Based Skills Assessment Battery (UPSA) | At baseline,2-week, 4-week, and 8-week follow-up.
Side-effects of tACS | At each stimulation session,up to 2 weeks.
The MATRICS Consensus Cognitive Battery (MCCB) | At 4-week and 8-week follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Chunbo Li, Ph.D., Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No